CLINICAL TRIAL: NCT00106301
Title: A Multicenter, Open-Label Continuation Trial Evaluating the Tolerability and Activity of FK228 in Patients That Have Completed a Prior Clinical Study With FK228
Brief Title: Continuation Trial Evaluating the Tolerability and Activity of FK228 in Patients That Completed Prior Study With FK228
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-228-0007
Record Dates: First submitted 2005-03-22; First posted 2005-03-23 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Renal Cell; Prostatic Neoplasms
Keywords: FK228; Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Prostatic Neoplasms | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FK228 (romidepsin) (Experimental): romidepsin
  Interventions: Drug: FK228 (romidepsin)

INTERVENTIONS:
Drug: FK228 (romidepsin) — Patients were continued at the same dose of romidepsin as in the previous study, which could have been 13 mg/m2 or a reduced dose of 10 mg/m2, administered intravenously over 4 hours on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: romidepsin

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of extended treatment with FK228 in patients with metastatic renal cell carcinoma or hormone refractory prostate cancer who have at least demonstrated stable disease on prior Fujisawa sponsored FK228 clinical trials.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized, open-label, single arm, continuation trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed 6 cycles of therapy in a prior Fujisawa-sponsored FK228 clinical trial;
* Patient has immediate past participation (not to exceed 21 days from Day 15 of cycle 6 in the previous study) in a prior Fujisawa-sponsored FK228 clinical trial;
* Patient has demonstrated stable disease, partial response or complete response as best overall response in their prior Fujisawa-sponsored FK228 clinical trial.

Exclusion Criteria:

* Patient has been on a prior Fujisawa-sponsored FK228 clinical trial, left the trial and then received alternative anti-neoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2006-09-01 (Actual); Study Completion 2006-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 6 months

SECONDARY OUTCOMES:
To evaluate the effect of depsipeptide therapy on performance status as measured by the Karnofsky score assessment | Up to 6 months
To evaluate the time to objective disease progression. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William McCulloch, MB, FRCP, Study Director — Gloucester Pharmaceuticals Inc.
Locations (5):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Seattle Cancer Care Alliance, Seattle, Washington
- Royal Marsden Hospital, Sutton, United Kingdom

REFERENCES:
- [Background] Moreno L, Casanova M, Chisholm JC, Berlanga P, Chastagner PB, Baruchel S, Amoroso L, Gallego Melcon S, Gerber NU, Bisogno G, Fagioli F, Geoerger B, Glade Bender JL, Aerts I, Bergeron C, Hingorani P, Elias I, Simcock M, Ferrara S, Le Bruchec Y, Slepetis R, Chen N, Vassal G. Phase I results of a phase I/II study of weekly nab-paclitaxel in paediatric patients with recurrent/refractory solid tumours: A collaboration with innovative therapies for children with cancer. Eur J Cancer. 2018 Sep;100:27-34. doi: 10.1016/j.ejca.2018.05.002. Epub 2018 Jun 21. PMID 29936064
- [Background] Wolchok J. Putting the Immunologic Brakes on Cancer. Cell. 2018 Nov 29;175(6):1452-1454. doi: 10.1016/j.cell.2018.11.006. PMID 30500529
- [Background] Mansfield AS, Jen J. Predicting Treatment Response Based on RNA Expression in Large Datasets. Clin Cancer Res. 2019 Mar 1;25(5):1443-1445. doi: 10.1158/1078-0432.CCR-18-2823. Epub 2018 Nov 16. PMID 30446588
- [Background] Pal SK, Forero-Torres A, Thompson JA, Morris JC, Chhabra S, Hoimes CJ, Vogelzang NJ, Boyd T, Bergerot PG, Adashek JJ, Li H, Yu X, Gartner EM, Carret AS, Smith DC. A phase 1 trial of SGN-CD70A in patients with CD70-positive, metastatic renal cell carcinoma. Cancer. 2019 Apr 1;125(7):1124-1132. doi: 10.1002/cncr.31912. Epub 2019 Jan 9. PMID 30624766